CLINICAL TRIAL: NCT03105778
Title: Point of Care Precision and Sample Comparison Study of Minicare BNP at Innsbruck Hospital - MI-BNP-CE04-AN2016
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Philips Handheld Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: HHDx-08698
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure
Keywords: BNP; IVD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples will be retained for future research purposes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: standard blood draw as part of routine and fingerprick for capillary sample — All blood sample collection methods are standard routine procedures. These patients usually have an indwelling cannula from which blood samples are drawn. So no additional venipuncture is performed according to this study. The finger prick sample - taken only for study purposes - might be accompanied by small pain at the fingertip. But this pain is usually of short duration and tolerated very well. No unanticipated adverse events are expected to occur in this study.

SUMMARY:
Part 1 (POC Precision):

Objective :

Demonstrate that the Minicare BNP (im)precision in hands of the user is within the expected range of the Minicare BNP (im)precision. Part 2 (sample comparison)

Primary objective :

Compare Minicare BNP values from capillary whole blood from finger stick with EDTA whole blood from venous puncture.

Secondary objective :

Compare Minicare BNP values from EDTA whole blood and plasma with Li- Heparin whole blood and plasma from venous puncture.

DETAILED DESCRIPTION:
Study Design Part 1 (POC precision) Two levels of BNP control samples (Thermofisher) will be tested during 5 days, with 5 replicates per day by three different users to assess precision of the Minicare BNP. The two different levels need to be tested on the same analyzer by the same user. For this study, six analyzers are made available, meaning that each user will test 2 analyzers. In parallel this testing will be done at Philips to establish the expected POC (im)precision. The two (im)precision values will be compared to each other. The precision study will also be used as a proficiency study that is normally requested prior to starting enrolment. Study Design Part 2 (sample comparison)

Part 2 (Sample comparison):

This study will be a prospective European single site study with at least 100 patient samples, taken from patients presenting at the cardiology ward and coronary care unit with suspected/ diagnosed heart failure (HF) or other cardiac diseases and thus suspected elevated BNP values. The blood sample will be collected near the patient by a trained healthcare professional of the study site.

When testing capillary whole blood, the blood will be collected by a finger stick according to the local SOP's of the study site. Directly (within 1 minute) after finger stick, the blood will be transferred with capillary transfer devices, one without ant-coagulant and one containing EDTA as anti-coagulant, to the BNP cartridge that is positioned in the Minicare I-20 analyzer. Testing will be done near the bedside of the patient. Two venous whole blood tubes will be collected; one containing Li-Heparin and the other containing EDTA as anti-coagulant. The venous whole blood will be collected in the specific tubes by a venous puncture according to the local SOP's of the study site. The EDTA venous whole blood will be transferred to the Minicare BNP by using a pipet and a transfer device. The Li-Heparin and EDTA venous whole blood sample should be tested within 2 hours (keep at room temperature) after the blood is taken (preferably as soon as possible after blood taking). Li-Heparin and EDTA venous whole blood can be tested at the ward by a trained healthcare professional or in the lab by a trained lab technician. The Li-Heparin and EDTA whole blood sample will be transferred to the lab and centrifuged and tested within 2 hours after the blood is taken. The Li-Heparin and EDTA plasma should be tested within 2 hours (keep at room temperature) after the blood is taken (preferably as soon as possible after blood taking). Li- Heparin and EDTA plasma samples might be tested in the lab, dependent on local routine.

All patient samples will be tested in singleton. The time that the blood is taken and tested will be recorded for each sample. Study will continue until at least 100 patient samples covering the predefined concentration range have valid measurements. Due to experience from previous sample comparison studies (Lab2Go) the site expects the necessity to test up to 200 patients to find 100 patients within the required BNP ranges. The Minicare BNP test results will not be used as part of the patient diagnosis but only for sample comparison purposes. Testing for both Part 1 and Part 2 will be done according to the Clinical Brochure for Minicare BNP.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older
* patients with suspected/ diagnosed heart failure (HF)
* signed informed consent form

Exclusion criteria:

* Patients younger than 18 years
* Patients requiring emergency treatment, those with cognitive impairment or inability to understand study information, and those unwilling or unable to provide written consent
* Patients already participated in this study
* Pregnant or breastfeeding women
* Patients with known Hepatitis B or C or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient samples from eligible patients with BNP requests, available at the test site
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
POC precision objective | June 2017
  Demonstrate that the Minicare BNP (im)precision in hands of the user is within the expected range of the Minicare BNP (im)precision.
Sample comparison objective | June 2017
  Compare Minicare BNP values from capillary whole blood from finger stick with EDTA whole blood from venous puncture.

SECONDARY OUTCOMES:
Sample comparison secondary objective | June 2017
  Compare Minicare BNP values from EDTA whole blood and plasma with Li- Heparin whole blood and plasma from venous puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Mair, Principal Investigator — Senior Staff member
Locations (1):
- Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Data outcome of study may be included in publication